CLINICAL TRIAL: NCT03836352
Title: A Phase 2, Open-label, Multicenter, Study of an Immunotherapeutic Treatment, DPX-Survivac in Combination With Low Dose Cyclophosphamide and Pembrolizumab, in Subjects With Selected Advanced and Recurrent Solid Tumours.
Brief Title: Study of an Immunotherapeutic, DPX-Survivac, in Combination With Low Dose Cyclophosphamide & Pembrolizumab, in Subjects With Selected Advanced & Recurrent Solid Tumors
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ImmunoVaccine Technologies, Inc. (IMV Inc.) (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P1719-SUR-Z11; Keynote 903 (Other: Sponsor)
Record Dates: First submitted 2019-02-07; First posted 2019-02-11 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Ovarian Cancer; Hepatocellular Carcinoma; Non-small Cell Lung Cancer; Bladder Cancer; Microsatellite Instability-High
Keywords: T cell activation; Immunotherapy; Ovarian; Hepatocellular Carcinoma; Non-small Cell Lung; Bladder; Microsatellite Instability-High; Survivin; Anti-PD-1; MK-3475
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Hepatocellular; Carcinoma, Non-Small-Cell Lung; Urinary Bladder Neoplasms | interventions — Cyclophosphamide; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (All cohorts) (Experimental): DPX-Survivac, Cyclophosphamide, Pembrolizumab
  Interventions: Other: DPX-Survivac; Drug: Cyclophosphamide; Drug: Pembrolizumab
- Arm 2 (Ovarian cohort only) (Experimental): DPX-Survivac, Pembrolizumab
  Interventions: Other: DPX-Survivac; Drug: Pembrolizumab

INTERVENTIONS:
Other: DPX-Survivac — SubQ injection (q9w)
Drug: Cyclophosphamide — PO (BID)
  Arms: Arm 1 (All cohorts)
Drug: Pembrolizumab — IV Infusion (q3w)
  Other Names: MK-3475

SUMMARY:
This study will assess the safety and efficacy of DPX-Survivac and low dose cyclophosphamide with pembrolizumab in subjects with selected advanced and recurrent solid tumours.

DETAILED DESCRIPTION:
This study is a Phase 2 with safety lead-in study to assess the safety and efficacy of DPX-Survivac, low dose cyclophosphamide, and pembrolizumab combination therapy in subjects with selected advanced and recurrent solid tumours. Two ovarian cancer arms will be recruited and randomized in this study, one with and one without cyclophosphamide. All other cohorts will be single arm, receiving treatment with the triple combination.

Up to 20 subjects, from any cohort, will be enrolled to assess the safety of study treatments before the study moves to the expansion phase. Once the safety lead-in is completed, the five cohorts will be expanded to recruit additional subjects following a Simon two stage design. Enrollment in the ovarian cancer cohort will be randomized 1:1 into two arms.

ELIGIBILITY:
Key Inclusion Criteria:

* Subjects with advanced or metastatic solid tumours who have completed treatment with first line therapy:

  1. Epithelial ovarian, fallopian tube, or peritoneal cancer
  2. Hepatocellular carcinoma
  3. Non-small cell lung cancer
  4. Urothelial cancer
  5. Microsatellite instability high solid tumours, other than the above indications
* Radiologic and/or biochemical evidence of disease progression
* Completion of pre-treatment tumour biopsy
* Must have measurable disease by RECIST v1.1
* Ambulatory with an ECOG 0-1
* Life expectancy ≥ 6 months
* Meet protocol-specified laboratory requirements

Key Exclusion Criteria:

* Chemotherapy or immunotherapy within treatment within 28 days of start of study treatment
* Radiotherapy within treatment within 2 weeks of start of study treatment
* Prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T cell receptor where subject was discontinued from that treatment due to a Grade 3 or higher immune-related toxicity
* For NSCLC subjects: Known EGFR mutations or ALK rearrangements
* Prior receipt of survivin-based vaccine(s) and/or immunotherapies
* Concurrent second malignancy other than non-melanoma skin cancer, cervical carcinoma in situ, or controlled bladder cancer
* Clinical ascites or pleural fluid that cannot be managed
* Malignant bowel obstruction or recent history of bowel obstruction
* For OvCa, subjects with any single lesion greater than 5 cm
* Autoimmune disease requiring treatment within the last two years (except replacement therapy)
* Recent history of thyroiditis
* Any history of (non-infectious) pneumonitis that required steroid therapy or current pneumonitis
* Presence of a serious acute or chronic infection
* Active CNS metastases and/or carcinomatous meningitis
* GI condition that might limit absorption of oral agents
* Allogenic tissue/solid organ transplant
* Other serious intercurrent chronic or acute illness, including myocardial infarction or cerebrovascular event within 6 months
* Ongoing treatment with steroid therapy or other immunosuppressive
* Receipt of live attenuated vaccines
* Acute or chronic skin and/or microvascular disorders
* Edema or lymphedema in the lower limbs > grade 2
* Severe hypersensitivity (≥ Grade 3) to pembrolizumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2018-12-21 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy as measured by objective response rate | Approximately 24 months
  Centrally evaluated using RECIST v1.1
Safety as measured by the rate of adverse events | Approximately 24 months
  Using the Common Terminology Criteria for Adverse Events (CTCAE) v5.0

SECONDARY OUTCOMES:
Objective response rate | Approximately 24 months
  Centrally evaluated using iRECIST
Duration of response | Approximately 24 months
Disease control rate | Approximately 24 months
Progression Free Survival | Approximately 24 months
Overall survival | Approximately 24 months

OTHER OUTCOMES:
Cell mediated immunology | Approximately 24 months
  As measured by antigen specific immune response in peripheral blood
Changes in immune cell infiltration | Approximately 24 months
  As measured by multiplex immunohistochemistry

CONTACTS AND LOCATIONS:
Locations (23):
- United States (15):
  - The University of Arizona Cancer Center, Tucson, Arizona
  - Cedars Sinai Medical Center: Samuel Oschin Comprehensive Cancer Center, Los Angeles, California
  - Boca Raton Regional Hospital, Lynn Cancer Institute, Boca Raton, Florida
  - Hematology Oncology Associates of the Treasure Coast, Port Saint Lucie, Florida
  - Comprehensive Hematology and Oncology, St. Petersburg, Florida
  - Winship Cancer Institute: The Emory Clinic, Atlanta, Georgia
  - James Brown Graham Cancer Center:University of Louisville Hospital, Louisville, Kentucky
  - Ochsner Cancer Institute, New Orleans, Louisiana
  - Allina Health, Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Christus St. Vincent Regional Cancer Center, Santa Fe, New Mexico
  - NYU Winthrop Hospital, Mineola, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of Toledo, Toledo, Ohio
  - Mary Crowley Cancer Research Center, Dallas, Texas
  - MD Anderson, Houston, Texas
- Canada (8):
  - William Osler Health System, Brampton, Ontario
  - Juravinski Cancer Center, Hamilton, Ontario
  - Southlake Regional Health Center, Newmarket, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Sunnybrook Research Institute, Toronto, Ontario
  - Centre hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec
  - McGill University Health Center, Montreal, Quebec
  - CHU de Québec-Université Laval, Québec, Quebec